CLINICAL TRIAL: NCT05379803
Title: A Single Arm, Multicenter Clinical Study of High-dose Furmonertinib in First-line Treatment of EGFR Mutated NSCLC With Central Nervous System (CNS) Metastases
Brief Title: High-dose Furmonertinib for First-line Treatment of EGFR Mutated NSCLC With Central Nervous System (CNS) Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORCE
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): furmonertinib 160 mg orally QD
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — furmonertinib 160 mg orally QD
  Other Names: AST2818

SUMMARY:
EGFR mutated NSCLC patiens with CNS metastases have poor prognosis. High-dose furmonertinib (160mg/day) have produced high CNS PFS and ORR in second-line for EGFR T790M mutated NSCLC. Whether EGFR mutated NSCLC with CNS metastases can benefit from first-line treatment of high-dose furmonertinib has not been reported. This study aims to investigate the efficacy and safety of high dose furmonertinib in first-line treatment of EGFR mutated NSCLC patiens.

DETAILED DESCRIPTION:
This is a single arm, multicenter clinical study and will recruit about 40 EGFR mutated NSCLC patients with CNS metastases in China. Furmonertinib is a third generation Epidermal Growth Factor Receptor (EGFR) tyrosine kinase inhibitor (TKI) .The recruited patients will receive high-dose furmonertinib (160mg/day) as first-line treatment. Whether EGFR mutated NSCLC with CNS metastases can benefit from first-line treatment of high-dose furmonertinib has not been reported. This study aims to investigate the efficacy and safety of high dose furmonertinib in first-line treatment of EGFR mutated NSCLC patiens.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any study-related procedure.
* Age ≥ 18 years.
* ECOG PS of 0 to 1 at screening,and with no clinically significant deterioration in the previous 2 weeks.
* Expected survival ≥12 weeks.
* Histologically or cytologically confirmed metastatic Non-Small Cell Lung Cancer (International Association for the Study of Lung Cancer and Joint Committee on the American Classification of Cancer, TNM Lung cancer stage 8). Documented validated results from local testing of either tumor tissue or blood confirming the presence of EGFR 19del or exon 21del L858R mutation. These mutations above may exist alone or together.
* According to RECIST 1.1, patients must have at least one central nervous system (CNS) metastatic tumor lesion at baseline that meets the following requirements: accurately and repeatably measurable at baseline, have no radiotherapy or biopsy.
* Patients who have untreated for advanced/metastatic non-small cell lung cancer, including chemotherapy, biological therapy, targeted therapy, immunotherapy, or experimental therapy, prior to initiation of study drug therapy. Patients who have received adjuvant therapy or neoadjuvant therapy (chemotherapy and/or radiotherapy) are allowed to enroll if there is no progression within 6 months of treatment. Patients who have received topical therapy (radiotherapy or perfusion therapy) are allowed to enroll if the lesion within the local therapeutic area is non-targeted.
* For premenopausal women with childbearing potential, a pregnancy test must be performed within 14 days before the first dose, and the pregnancy test (blood or urine test) must be negative; female subjects must not be lactating;
* Willing to use contraception.
* Voluntary and agree to follow the study treatment protocol as well as follow-up plan, and can accept the oral medicine treatment.

Exclusion Criteria:

* Small cell lung carcinoma;
* History of hypersensitivity to active or inactive excipients of investigational agent with a similar chemical structure.
* Confirmed EGFR 20 exon insertion mutations at any time after the initial diagnosis.
* Patient who receive prior treatment including any of the following:
* Any Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI).
* The patients who have received intrapleural perfusion therapy can only be enrolled 28 days or more after the pleural effusion is stable;
* Major surgery within 4 weeks of the first dose of investigational agent.
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of investigational agent;
* CYP3A4 strong inhibitor or strong inducer is used within 7 days prior to the first dose, or need to receive these drugs during the study period.
* Traditional Chinese medicine and traditional Chinese medicine preparations with anti-tumor as indications and with adjuvant treatment of tumor is used within 7 days prior to the first dose, or need to receive these drugs during the study period.
* Patients who are receiving drugs known to prolong QTc interval or may cause torsade de pointe and need to continue to receive these drugs during the study period.
* The time from the treatment with any other investigational product or its analogue to the first dose does not exceed 5 half-lives of the drug or 14 days, whichever is longer.
* Prior treatment with any systemic anti-cancer therapy for advanced Non-Small Cell Lung Cancer (NSCLC) including chemotherapy, biologic therapy, target therapy, immunotherapy, or any investigational drug, except neoadjuvant or adjuvant therapy before 6 months prior to the first dose investigational treatment.
* At the beginning of study treatment, any unresolved toxic reaction to prior treatment is present, which exceeds Grade 1 in accordance with Common Terminology Criteria for Adverse Events (CTCAE) (except for alopecia), and exceeds Grade 2 for prior platinum treatment-related neuropathy.
* Spinal cord compression; symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids.
* Diagnosed other malignant tumors or had a history of other malignant tumors in last 5 years, except for skin basal cell carcinoma, cervical carcinoma in situ and breast ductal carcinoma in situ which have been effectively controlled;
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of investigational agent.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, and active infection, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial.
* Past medical history of Interstitial Lung Disease (ILD), drug-induced Interstitial Lung Disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active Interstitial Lung Disease.
* Any evidence of corneal injury:
* Inadequate bone marrow reserve or organ function.
* QT prolongation or any clinically important abnormalities in rhythm and heart function.
* Patients who may have poor compliance with the research procedures and requirements, etc., as judged by investigators.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | The primary analysis of Progression-free survival (PFS) based on investigator assessment will occur when PFS maturity is observed at approximately 26 months after the first patient begin study treatment
  Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression.

SECONDARY OUTCOMES:
Central nervous system (CNS) progression-free survival | Central nervous system (CNS) progression-free survival (PFS) analysis based on investigator assessment will occur at approximately 26 months after the first patient begin study treatment.
  CNS PFS is defined as the time from beginning of study treatment until the date of objective progression of central nervous system or death (by any cause in the absence of CNS progression), regardless of whether the patient withdraws from study treatment or receives another anti-cancer therapy prior to progression.
Objective Response Rate | Objective Response Rate analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 26 months from the first patient begin study treatment.
  defined as the number (%) of patients with response of Complete Response or Partial Response.
Disease Control Rate | Disease Control Rate analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 26 months from the first patient begin study treatment.
  defined as the number (%) of patients with CNS lesion response of Complete Response or Partial Response.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China